CLINICAL TRIAL: NCT02286596
Title: Comparisons of Two Low-density Lipoprotein Apheresis Systems in Patients With Homozygous Familial Hypercholesterolemia
Acronym: APHERESE
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, MD, PhD, FRCP, Laval University
Other Study IDs: APHERESE
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- heparin-induced extracorporeal LDL precipitation: Lipid apheresis treatment for 3 hours
  Interventions: Device: heparin-induced extracorporeal LDL precipitation
- dextran sulfate adsorption: Lipid apheresis treatment for 3 hours
  Interventions: Device: dextran sulfate adsorption

INTERVENTIONS:
Device: heparin-induced extracorporeal LDL precipitation — Lipid apheresis for 3 hours
  Other Names: Futura
  Groups: heparin-induced extracorporeal LDL precipitation
Device: dextran sulfate adsorption — Lipid apheresis for 3 hours
  Other Names: Kaneka
  Groups: dextran sulfate adsorption

SUMMARY:
Homozygous familial hypercholesterolemia (HoFH) is characterized by a six- to eight-fold raise in plasma LDL-cholesterol (LDL-C) concentrations and atherosclerotic coronary artery disease usually occur before the age of 20 if untreated. Lipid apheresis (LA) has been proved to be a reliable method to decrease LDL-C concentrations and therefore decrease cardiovascular disease risk in HoFH. The objective of this crossover study was to compare efficacy of LA performed with heparin-induced extracorporeal LDL precipitation to dextran sulfate adsorption on the reduction of lipids, inflammatory markers, adhesion molecules and LDL particles size in a cohort of HoFH subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-65 years
* Subjects with homozygous familial hypercholesterolemia:
* Carrier of a mutation in the LDL receptor gene

Exclusion Criteria:

* Subjects with a previous history of cardiovascular disease
* Subjects with Type 2 diabetes
* Were pregnant or nursing;
* Subjects with a history of cancer
* Subjects with acute liver disease, hepatic dysfunction, or persistent elevations of serum transaminases
* Subjects with a secondary hyperlipidemia due to any cause
* History of alcohol or drug abuse within the past 2 years
* hormonal treatment
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with homozygous familial hypercholesterolemia already treated with LDL apheresis using both systems being compared (HELP vs Dextran)
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in plasma lipid levels between the two lipid apheresis treatment | At the end of the two lipid apheresis (Week 0 and 2)

SECONDARY OUTCOMES:
Change in plasma adhesion molecule levels between the two lipid apheresis treatment | At the end of the two lipid apheresis (Week 0 and 2)
Change in plasma inflammatory marker levels between the two lipid apheresis treatment | At the end of the two lipid apheresis (Week 0 and 2)
Change in LDL particle size between the two lipid apheresis treatment | At the end of the two lipid apheresis (Week 0 and 2)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada